CLINICAL TRIAL: NCT01303276
Title: Retinal Blood Flow in Response to an Intravitreal Injection of Ranibizumab for Central Retinal Vein Occlusion
Brief Title: Retinal Blood Flow in Response to an Intravitreal Injection of Ranibizumab for Central Retinal Vein Occlusion (CRVO)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Christopher Hudson, University of Toronto
Other Study IDs: CRVO-blood flow study
Record Dates: First submitted 2011-02-15; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Central Retinal Vein Occlusion
Keywords: retinal vein occlusion; anti-VEGF; blood flow
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anti-VEGF group: Patients who are clinically indicated for the intravitreal injection of ranibizumab
- Age-matched controls: Group of healthy participants who will be age and gender matched

SUMMARY:
Ranibizumab (Lucentis, Genentech) is an off-label drug used for the clinical treatment of central retinal vein occlusion, which is one of the most common retinal vascular disorders. Despite its clinical effectiveness, concerns remain regarding the systemic effects of the drug and previous studies have noted retinal arteriolar vasoconstriction following a ranibizumab injection. We aim to provide a physiological basis to these observations by assessing retinal blood flow before and after the ranibizumab injections. Specifically, we will assess the blood flow parameters (i.e. retinal vessel diameter, velocity & flow) immediately before the first injection and post-injection over a follow-up continued treatment period.

DETAILED DESCRIPTION:
Ranibizumab is an antibody fragment designed to inhibit the activity of Vascular Endothelial Growth Factor (VEGF), which is responsible for the neovascularization and retinal edema responsible for interference of normal vision in central retinal vein occlusion. However, VEGF has a role in the vasculature as a vasodilator where it alters the expression of tight junction proteins and upregulates the release of the vasodilator nitric oxide. Consequently, intravitreal ranibizumab injections could result in systemic inhibition of VEGF, leading to long-term retinal arteriolar vasoconstriction and potentially adverse cerebrovascular and myocardial accidents. Therefore, evaluating retinal blood flow would provide a physiological foundation to this concern and provide physicians with valuable information regarding the risks of continued ranibizumab therapy.

Given the role of VEGF as a vasodilator in the vasculature where it works to alter the expression of tight junction proteins and the production of vasoactive substances especially nitric oxide, inhibiting this molecule with ranibizumab could result in vasoconstriction in these vessels. We hypothesize that vasoconstriction and decreased retinal blood flow will be observed after an intravitreal injection of ranibizumab for treatment of central retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* central retinal vein occlusion scheduled for first intravitreal injection of ranibizumab as part of their clinical care

Exclusion Criteria:

* previous history of intravitreal therapy,
* history of thromboembolic events,
* glaucoma or an intraocular pressure >21 mmHg
* diabetes mellitus or altered blood viscosity syndromes
* blood donation in the previous 2 weeks
* refractive error of +/- 6.00 DS and/or 2.00 DC

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with central retinal vein occlusion will be recruited from the Retina Clinics of Toronto Western Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Quantitative change in retinal blood flow | Baseline, 7, 30 days
  Retinal blood flow will be measured using Canon Laser Blood Flowmeter

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (LogMAR, EDTRS) | Baseline, 7, 30 days
  Best Corrected Visual Acuity will be examined using 96% and 10 % contrast EDTRS letter charts

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hudson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada